CLINICAL TRIAL: NCT02608879
Title: Oral Care Protocol for the Management of Chemotherapy and Radiation Therapy-Induced Oral Mucositis
Acronym: OMDP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14-00082
Record Dates: First submitted 2015-11-13; First posted 2015-11-20 (Estimated); Results first posted 2020-08-28 (Actual); Last update posted 2020-08-28 (Actual); Status verified 2020-08

CONDITIONS: Oral Mucositis; Oral Cancer
Keywords: proinflammatory cytokines; microbiome; radiation therapy
MeSH Terms: conditions — Stomatitis; Mouth Neoplasms | interventions — Periodontal Debridement; Dental Scaling; High-Energy Shock Waves; Chlorhexidine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- OMDP Group (Experimental): Subjects randomized to this group will attend weekly visits and receive a full dental cleaning, as well as have their gums/tongue cleaned by a dental professional. Subjects will also receive standard of care oral hygiene instructions.
  Interventions: Procedure: Oral Mucosa Deterging and Periodontal Debridement (OMDP); Procedure: Dental scaling, ultrasonic; Other: Chlorhexidine
- Control Group (Other): Subjects assigned to the control group will receive standard of care oral health instructions and will come for bi-weekly treatment visits where they will have their teeth cleaned (brushed) by a dental professional.
  Interventions: Procedure: Standard of Care Oral Hygiene Instructions

INTERVENTIONS:
Procedure: Oral Mucosa Deterging and Periodontal Debridement (OMDP) — OMDP consists of a regimen of frequent professional oral prophylaxis including tooth cleaning, tooth polishing and flossing, and the cleaning of the periodontum and oral mucosa. This is an intervention that is implemented prior to and maintained throughout the entire cycle of the radiation or chemoradiation.
  Arms: OMDP Group
Procedure: Standard of Care Oral Hygiene Instructions — Subjects assigned to this intervention will receive standard of care oral hygiene instructions, including in-person instruction and materials to reference at home. Subjects will also have their teeth brushed and flossed bi-weekly by a dental professional.
  Arms: Control Group
Procedure: Dental scaling, ultrasonic — An ultrasonic dental scaler will be used to clean the teeth
  Arms: OMDP Group
Other: Chlorhexidine — Non-alcoholic chlorhexidine will be used as part of the OMDP protocol
  Arms: OMDP Group

SUMMARY:
The purpose of this study is to determine the effects of a novel oral care protocol on the severity and pain of oral mucositis in patients receiving radiation and/or chemotherapy for head and neck cancers. The secondary objectives are to characterize the microbiome associated with oral mucositis, measure salivary proinflammatory cytokines, and evaluate other clinical indicators of the intervention. Participants will be enrolled prior to beginning radiation and/or chemotherapy, and will be randomized to receive either the oral health protocol or standard of care oral hygiene.

DETAILED DESCRIPTION:
Oral mucositis (OM) is one of the most debilitating adverse effects in cancer patients treated with chemotherapy or radiation (RT). Currently, there are no effective therapies or prevention for mucositis, while several clinical studies have suggested that professional oral care could effectively reduce the severity of Radiation Therapy or chemotherapy-induced oral mucositis. Palliative treatment, rather than preventive or curative measures, remains the standard of care. Evidence-based guidelines do not provide consistent recommendations for the prevention, treatment and management of oral mucositis.

The investigators hypothesize that a monitored regimen of professional oral hygiene prevents harmful ecological shifts in the oral cavity, improve oral health and reduce the duration and severity of Oral Mucositis in cancer patients, consequently improving their overall quality of life during treatment. Moreover, the investigators hypothesize that the weekly oral hygiene regimen performed by an oral health professional is more effective in treating and preventing mucositis than current standard-of-care treatments.

The principal investigator of this project has developed a novel oral care regimen protocol for the treatment of oral mucositis. The "Oral Mucosa Deterging and Periodontal Debridement" (OMDP) protocol consists of a regimen of frequent professional oral prophylaxis including tooth cleaning, tooth polishing and flossing, and the debridement of the periodontium and deterging of the oral mucosa. This is an intervention that is implemented prior to and maintained throughout the entire cycle of the radiation or chemoradiation. Co-adjuvant treatments such as intense fluoride treatments, oral hygiene instructions and palliative mouth-rinses are also part of the protocol. The hypothesis is that repeated professional prophylaxis of the oral cavity would protect the healthy oral tissue against infection and inflammation often associated with severe cases of mucositis, and consequently reduces mucositis incidence and duration.

Participants in this study would attend approximately 9 study visits over the course of 16-18 weeks, depending on their specific cancer treatment plan. Study participants will be randomized to receive either the oral health protocol, which they will receive on a weekly basis, or standard of care oral hygiene instructions and tooth brushing, preformed on a bi-weekly basis.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patient aged 18 years or older;
2. Patients must sign an informed consent before data collection, screening, or initiation of study procedures;
3. Patients who are scheduled to undergo radiation or chemoradiation treatment for head/neck cancer;
4. Patients who have a minimum of 6 natural teeth at the time of enrollment.

Exclusion Criteria:

1. Female patients who are pregnant or lactating at the baseline/screening visit;
2. Patient participating in another biomedical/oral health research study that would interfere with participating in this study;
3. Patient deprived of freedom, under supervision or guardianship;
4. Patient unable to attend to scheduled medical monitoring due to geographical, social or mental reasons;
5. Immune compromised or other serious medical conditions, regardless of whether the condition is controlled or not;
6. Patient who requires pre-medication prior to dental treatment;
7. Any patient, in the opinion of the Investigator, who is unable or unlikely to comply fully with the study requirements or procedures for any reason (e.g. major surgical resection of intra-oral structures which would prevent oral care intervention, edentulous, severe periodontal disease, etc).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2014-03; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Corby, DDS, MS, Principal Investigator — NYU Langone Medical Center
Locations (1):
- NYU Langone Medical Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Not Randomized: Subjects in this study were randomized at the time oral mucositis (OM) was developed (approximately week 2-4). Subjects who met inclusion criteria at the time of enrollment, but did not meet continuation criteria at the time OM was developed were not randomized and were dropped from the study.
Period: Overall Study
Arm/Group | OMDP Group | Control Group | Not Randomized
Started | 10 | 6 | 3
Completed | 9 | 6 | 0
Not Completed | 1 | 0 | 3
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Did not meet continuation criteria | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | OMDP Group | Control Group | Not Randomized | Total
Number analyzed (Participants) | 10 | 6 | 3 | 19
Age, Continuous [Mean (Full Range); unit: years] | 55.8 [30 to 79] | 55.5 [48 to 64] | 67.33 [50 to 77] | 57.5 [30 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 1 | 7
  Male | 6 | 4 | 2 | 12
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaskan | 0 | 1 | 0 | 1
  Asian or Pacific Islander | 1 | 0 | 0 | 1
  Black, not of Hispanic-American Origin | 1 | 1 | 0 | 2
  Hispanic-American | 1 | 0 | 0 | 1
  White, not of Hispanic-American Origin | 6 | 4 | 1 | 11
  Other/Unknown | 1 | 0 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Oral Mucositis Severity - WHO Scale
Description: OM severity will be assessed by the WHO Oral Mucositis Scale at each follow-up visit.
  The WHO Oral Mucositis Scale is a 5 point scale (0 to 4) with the following scoring system:
  0=None
  1. Soreness with erythema
  2. Erythema, ulcers, can eat solids
  3. Ulcers, liquid diet only
  4. Alimentation not possible
Time Frame: End of Radiation Treatment (approximately week 7)
Population: Data from the one participant in the OMDP group who was lost to follow up was not analyzed for this measure.
Measure: Number; unit: participants
Arm/Group | OMDP Group | Control Group
Number analyzed (Participants) | 9 | 6
participants
  WHO score of 0 | 3 | 3
  WHO score of 1 | 0 | 0
  WHO score of 2 | 6 | 2
  WHO score of 3 | 0 | 0
  WHO score of 4 | 0 | 1

2. Primary Outcome: Oral Mucositis Severity - NCI Scale
Description: OM severity will be assessed by the NCI-CTCAE Scale (National Cancer Institute - Common Toxicity Criteria and Grading of Adverse Events) at each follow-up visit.
  The NCI-CTCAE is a 5 point scale (1-5) with the following grading system:
  1. Erythema of the mucosa
  2. Patchy ulcerations or pseudomembranes
  3. Confluent ulcerations or pseudomembranes; bleeding with minor trauma
  4. Tissue necrosis; significant spontaneous bleeding; life-threatening consequences
  5. Death
Time Frame: End of Radiation Treatment (approximately week 7)
Population: Data from the one participant in the OMDP group who was lost to follow up was not analyzed for this measure.
Measure: Number; unit: participants
Arm/Group | OMDP Group | Control Group
Number analyzed (Participants) | 9 | 6
participants
  CTCAE score of 1 | 6 | 3
  CTCAE score of 2 | 2 | 1
  CTCAE score of 3 | 1 | 2
  CTCAE score of 4 | 0 | 0
  CTCAE score of 5 | 0 | 0

3. Secondary Outcome: Level of Oral Pain (FACES Scale)
Description: The FACES Scale is a 6 point scale which ranges from 0-10 (and includes even numbers only). The scale is accompanied by illustrations of faces which represent each score. The subjects is shown the scale and asked to choose the face that best depicts the pain they are experiencing.
  0=No hurt 2=Hurts a little bit 4=Hurts a little more 6=Hurts even more 8=Hurts a whole lot 10-Hurts the worst you could imagine
Time Frame: End of Radiation Treatment (approximately week 7)
Population: Data from the one participant in the OMDP group who was lost to follow up was not analyzed for this measure.
Measure: Number; unit: participants
Arm/Group | OMDP Group | Control Group
Number analyzed (Participants) | 9 | 6
participants
  FACES score of 0 | 0 | 1
  FACES score of 2 | 6 | 3
  FACES score of 4 | 1 | 1
  FACES score of 6 | 1 | 1
  FACES score of 8 | 1 | 0
  FACES score of 10 | 0 | 0

4. Secondary Outcome: Mean Difference in the Relative Abundance of Oral Microbial Species of the Cheek (Right Side) From Baseline to Onset of Oral Mucositis
Description: The number of each type of microbial species will be quantified and compared at each follow-up visit. Relative abundance for each species will be measured and reported. Relative abundance is a measure of the proportion of an organism of a particular kind (in this case, each microbial species) relative to the total number of organisms (the other microbial species) in the area.
  A positive mean value indicates that the species was present in greater quantities at baseline. A negative mean value indicates that the species was present in greater quantities at onset of oral mucositis.
  For this data, the top five most abundant microbial species are presented.
Time Frame: Baseline to Onset of Oral Mucositis
Population: Data were only collected for the OMDP Grouip because they are the only group that developed oral mucositis.
Measure: Mean (95% Confidence Interval); unit: Proportion of oral microbial species
Arm/Group | OMDP Group
Number analyzed (Participants) | 9
Proportion of oral microbial species
  Stomatobaculum sp oral taxon 97 | 2.6517 [0.7038302 to 4.5995841]
  Leptotrichia sp oral taxon | 1.8354 [0.1348964 to 3.5358455]
  Haemophillus Genus probe 3 | -2.2123 [-4.2835766 to -0.1410081]
  Veillonella Genus probe 2 | -0.9269246 [-1.8325844 to -0.0212649]
  Gemella Haemolysans | -0.7559120 [-1.6171195 to 0.1052956]

5. Secondary Outcome: Mean Difference in the Relative Abundance of Oral Microbial Species of the Cheek (Left Side) From Baseline to Onset of Oral Mucositis
Description: as for outcome 4
Time Frame: Baseline to Onset of Oral Mucositis
Population: This outcome measure was only collected in the OMDP Group because this is the only arm where participants developed Oral Mucositis.
  Two subjects were excluded from this analysis due to a diagnosis of HIV, which the investigator determined would alter the microbial makeup of the oral cavity.
Measure: Mean (95% Confidence Interval); unit: Proportion of oral microbial species
Arm/Group | OMDP Group
Number analyzed (Participants) | 9
Proportion of oral microbial species
  Fusobacterium periodonticum | 2.3367705 [0.5610779 to 4.1124631]
  Leptotrichia sp oral taxon 417 | 1.7988509 [0.3998338 to 3.19778681]
  Stomatobaculum sp oral taxon 97 | 2.5104787 [0.4810140 to 4.5399434]
  Gemella Haemolysans | -0.6947840 [-1.6371024 to 0.2475345]
  Prevotella histicolla | -0.8316186 [-2.0134734 to 0.3502363]

6. Secondary Outcome: Mean Difference in the Relative Abundance of Oral Microbial Species of the Tongue (Right Side) From Baseline to Onset of Oral Mucositis
Description: as for outcome 4
Time Frame: Baseline to Onset of Oral Mucositis
Population: as for outcome 5
Measure: Mean (95% Confidence Interval); unit: Proportion of oral microbial species
Arm/Group | OMDP Group
Number analyzed (Participants) | 9
Proportion of oral microbial species
  Haemophillus Genus probe 3 | -3.545091 [-4.9414618 to -2.1487203]
  Gemella Haemolysans | -2.1439002 [-3.2226984 to -1.0651020]
  Streptococcus Genus probe 1 | -0.9359749 [-1.5210515 to -0.3508983]
  Leptotrichia sp oral taxon 417 | 1.3618774 [0.3917063 to 2.3320485]
  Gemella Sanguinis | 2.9317234 [0.8166947 to 4.8467521]

7. Secondary Outcome: Mean Difference in the Relative Abundance of Oral Microbial Species of the Tongue (Left Side) From Baseline to Onset of Oral Mucositis
Description: as for outcome 4
Time Frame: Baseline to Onset of Oral Mucositis
Population: as for outcome 5
Measure: Mean (95% Confidence Interval); unit: Proportion of oral microbial species
Arm/Group | OMDP Group
Number analyzed (Participants) | 9
Proportion of oral microbial species
  Gemella Sanguinis | 3.1061673 [1.6923225 to 4.500120]
  Stomatobaculum sp oral taxon 97 | 3.6522501 [1.9517525 to 5.3527476]
  Fusobacterium periodonticum | 2.8036767 [1.3181513 to 4.2892021]
  Gemella Haemolysans | -1.5662996 [-2.4326884 to -0.6999108]
  Haemophillus Genus probe 3 | -2.9178458 [-4.6320329 to -1.2036587]

8. Secondary Outcome: Change in the Level of Salivary Proinflammatory Cytokines From Baseline to 16 Weeks
Description: The level of salivary proinflammatory cytokines will be compared between the two groups at each follow-up visit.
Time Frame: Baseline and 16 weeks (final study visit)
Population: Due to financial limitations, not all data could be analyzed at this time. Samples were collected and may be analyzed at a later point. Analyzed samples were limited to those collected from subjects with oropharyngeal cancer (i.e. samples from subjects with cancer of the oral cavity were not analyzed at this time).
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | OMDP Group | Control Group
Number analyzed (Participants) | 5 | 5
pg/mL
  IFN-ɣ | -0.7228 (0.18) | 0.5782 (0.5782)
  IL-1 | -0.7184 (0.3918) | 0.5747 (0.5747)
  IL-10 | -0.4503 (0.0823) | 0.3603 (0.3603)
  IL-12p70 | -0.4503 (0.0823) | 0.3603 (0.3603)
  IL-13 | -0.8873 (0.2511) | 0.7099 (0.7099)
  IL-2 | -0.2754 (0.0142) | 0.2203 (0.2203)
  IL-4 | -0.3639 (1.3222) | 0.2911 (0.2911)
  IL-6 | -0.5358 (0.9856) | 0.4286 (0.4286)
  IL-8 | -0.7407 (0.2868) | 0.5925 (0.5925)
  TNF-α | -0.5881 (0.0627) | 0.4705 (0.4705)

9. Secondary Outcome: Change in Quality of Life as Measured by the Composite Score of the EORTC
Description: Quality of life will be measured using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC) and Head & Neck module (EORTC-H&N) and compared between the two groups at each follow-up visit.
  There is not a single composite score for the entire questionnaire, but rather composite scores for each type of assessment (e.g. physical functioning, global health, swallowing, etc.). Possible scores range from 0-100. A lower score indicates low levels of that trait, which a higher score indicates high levels of that trait (e.g. a 100 for "physical functioning" indicates a high level of physical function).
Time Frame: Baseline to the peak of mucositis (approximately week 4)
Population: Only data from subjects with oropharyngeal cancer were included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | OMDP Group | Control Group
Number analyzed (Participants) | 5 | 5
units on a scale
  Physical Functioning Score | 11.7 (8.4) | -3.9 (6.1)
  Global Health Status | -20.9 (16) | -3.4 (7.3)
  H&N Swallowing Scale | 2 (23.1) | -10 (22.1)

ADVERSE EVENTS:
Arm/Group | OMDP Group | Control Group | Not Randomized
Serious Adverse Events (participants affected / at risk) | 1/10 | 0/6 | 1/3
Other Adverse Events (participants affected / at risk) | 10/10 | 6/6 | 2/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OMDP Group (N=10) | Control Group (N=6) | Not Randomized (N=3)
Abnormal liver function (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OMDP Group (N=10) | Control Group (N=6) | Not Randomized (N=3)
Oral Mucositis (Gastrointestinal disorders) | 10 | 6 | 2
Allergic reaction (General disorders) | 1 | 1 | 0
Candidiasis (Infections and infestations) | 5 | 2 | 1
Dry Mouth/throat (Gastrointestinal disorders) | 7 | 5 | 0
Sore throat (Gastrointestinal disorders) | 1 | 3 | 0
Nausea (Gastrointestinal disorders) | 7 | 3 | 0
Dehydration (General disorders) | 1 | 0 | 0
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Cacogeusia (Gastrointestinal disorders) | 0 | 1 | 0
Edema (Blood and lymphatic system disorders) | 1 | 0 | 0
Lymphoedema (Blood and lymphatic system disorders) | 0 | 1 | 0
Dysgeusia (Gastrointestinal disorders) | 1 | 1 | 0
Radiation dermatitis (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Fatigue (General disorders) | 0 | 1 | 1
Shingles (Infections and infestations) | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0
Hearing loss (Ear and labyrinth disorders) | 1 | 0 | 0
Cold/flu (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Chemotherapy induced rash (Surgical and medical procedures) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Hiccups with acid reflux (Gastrointestinal disorders) | 1 | 0 | 0
Heartburn (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Shoulder pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Hypogeusia (Gastrointestinal disorders) | 1 | 0 | 0
Burning on the tongue (Gastrointestinal disorders) | 1 | 0 | 0
Herpetic lesion (Infections and infestations) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes